CLINICAL TRIAL: NCT00523666
Title: Diffusion Tensor Weighted MRI in Alzheimer's Disease: Prediction and Mapping of Symptomatic and Disease Modifying Treatment Effects of Galantamine (Reminyl®)
Brief Title: Diffusion Tensor Weighted MRI in Alzheimer's Disease Modifying Treatment Effects of Galantamine (Reminyl®)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DTI001; EudraCT 2005-003762-41
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; diffusion tensor imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Galantamine (Reminyl®)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo/Galantamine (Reminyl®)

INTERVENTIONS:
Drug: Galantamine (Reminyl®) — 8mg - 24mg
  Arms: 1
Drug: Placebo/Galantamine (Reminyl®) — Patients are treated double-blind with placebo for 6 months, followed by treatment with Galantamine (Reminyl®) for another 6 months.
  Dose scheme: 8mg-24mg
  Arms: 2

SUMMARY:
Alzheimer's disease (AD) is characterized by progressive subcortical and cortical neuronal degeneration. AD patients differ in the time course of neuronal degeneration and accompanying cognitive decline.

With recent advances in MR imaging, including optimized data acquisition and processing techniques, tools that are especially well suited for tracking long-term pathological changes as well as drug treatment effects have become available. In addition to structural imaging, new acquisition and analysis techniques have been developed to determine integrity of subcortical fiber tracts in vivo.

In the present project we propose to determine predictors of disease progression and treatment response and investigate potential treatment effects on structural disease progression, covering the continuum from axonal degeneration to cortical neuronal loss taking advantage of recent advances in MRI acquisition and analysis techniques.

DETAILED DESCRIPTION:
The outlined project will provide data to determine the value of cortical and subcortical volumetric and diffusion markers of neuronal degeneration to predict disease progression and response to (acetyl-)cholinergic treatment with Galantamine (Reminyl®). Furthermore, analysis of longitudinal MRI data in respect to cortical and subcortical atrophy and fiber degeneration will provide an estimate of the potential of new MRI analysis techniques to determine effects of (acetyl-)cholinergic treatment on rates of disease progression. Finally, the proposed study will allow determining the potential value of a new MRI technique, diffusion tensor imaging, to show the morphological correlate of cortical disconnection in AD and to map progression and treatment related effects on subcortical fiber tract integrity in AD.

The major scientific value of this project is the combined description of the effect of Galantamine (Reminyl®) on disease progression on the structural level of analysis in AD. The data from this project may help to identify predictors of treatment response and to elucidate the mechanisms of drug action of Galantamine (Reminyl®) in AD.

ELIGIBILITY:
Inclusion Criteria:

* male of female patients aged ≥ 55years, fulfilling criteria of the National Institute of Neurological and Communicative Disease and Stroke (NINCDS) and the Alzheimer's Disease and Related Disorders Association (ADRDA) for the diagnosis of clinically probable AD
* MMSE score > 16
* no evidence for other psychiatric axis I disorders according to DSM- IV criteria
* no evidence for cerebrovascular disease (radiological confirmed), cardiac or cerebral infarct (three months before the study), thyroid disease and other neurodegenerative or neuroinflammatory disorders. No evidence for acute or unstable medical condition.
* no risk factors of hypertension, cardiac disease (e.g. angina pectoris, congestive heart failure, right bundle branch block, or arrhythmias), diabetes mellitus (stable within 3 months)
* no history of drug/alcohol abuse
* no history of panic attacks or claustrophobia (due to requirements of the MRI examinination)
* no surgical implants or non-fixed metallic particles
* patient has not taken a previously approved cholinesterase inhibitor or memantine, which has been discontinued at least 6 weeks prior to the Screening
* patient is able to provide written Informed Consent to participate study. If, at investigator's discretion, a patient is considered not to be capable to give legal consent, then written consent must also be obtained from the patient's legally acceptable representative.

Exclusion Criteria:

* no evidence of memory or other cognitive impairments, verified by clinical history and cognitive testing
* previous or current history of degenerative or ischemic disorders of the peripheral or central nervous system
* previous or current history of systemic disorders
* no ability to participate and no willing to give informed consent and comply with the study restrictions
* MMSE score < 16 range

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-09; Study Completion 2008-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Hampel, MD, Study Director — Dementia Research Section and Memory Clinic, Department of Psychiatry, Nussbaumstrasse 7, 80336 Munich, Germany; Stefan Teipel, MD, Principal Investigator — Dementia Research Section and Memory Clinic, Department of Psychiatry, Nussbaumstrasse 7, 80336 Munich, Germany
Locations (1):
- Ludwig-Maximilian University of Munich, Munich, Germany

REFERENCES:
- [Background] Teipel SJ, Stahl R, Dietrich O, Schoenberg SO, Perneczky R, Bokde AL, Reiser MF, Moller HJ, Hampel H. Multivariate network analysis of fiber tract integrity in Alzheimer's disease. Neuroimage. 2007 Feb 1;34(3):985-95. doi: 10.1016/j.neuroimage.2006.07.047. Epub 2006 Dec 12. PMID 17166745
- [Background] Sydykova D, Stahl R, Dietrich O, Ewers M, Reiser MF, Schoenberg SO, Moller HJ, Hampel H, Teipel SJ. Fiber connections between the cerebral cortex and the corpus callosum in Alzheimer's disease: a diffusion tensor imaging and voxel-based morphometry study. Cereb Cortex. 2007 Oct;17(10):2276-82. doi: 10.1093/cercor/bhl136. Epub 2006 Dec 12. PMID 17164468
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] Blautzik J, Keeser D, Paolini M, Kirsch V, Berman A, Coates U, Reiser M, Teipel SJ, Meindl T. Functional connectivity increase in the default-mode network of patients with Alzheimer's disease after long-term treatment with Galantamine. Eur Neuropsychopharmacol. 2016 Mar;26(3):602-13. doi: 10.1016/j.euroneuro.2015.12.006. Epub 2015 Dec 10. PMID 26796681